CLINICAL TRIAL: NCT00434499
Title: An Exploratory Study to Evaluate the Ability of Epigallocatechin Gallate to Simultaneously Improve Metabolic and Cardiovascular Actions of Insulin in Healthy and Obese Subjects
Brief Title: Effect of EGCG on the Body's Response to Insulin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not funded
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kashif Munir, Assistant Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00048859
Record Dates: First submitted 2007-02-10; First posted 2007-02-13 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Hypertension; Obesity; Type 2 Diabetes; Insulin Resistance
Keywords: Green Tea; Insulin Resistance; Endothelial Dysfunction; Nitric Oxide; Inflammation; Obesity; Overweight; Diabetes Type 2; High Blood Pressure; Healthy Volunteer; HV
MeSH Terms: conditions — Hypertension; Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo first (Active Comparator): placebo first then crossover to EGCG
  Interventions: Drug: EGCG
- EGCG first (Active Comparator): EGCG first then crossover to placebo
  Interventions: Drug: EGCG

INTERVENTIONS:
Drug: EGCG — EGCG 400 mg by mouth twice/daily for 4 weeks duration.

SUMMARY:
This study will examine whether epigallocatechin gallate (EGCG), a major component of green tea, affects how the body responds to insulin in healthy and obese people. Insulin is not as effective in people who are overweight, have high blood pressure or diabetes. This condition is known as insulin resistance. Laboratory studies suggest that green tea or EGCG treatment lowers blood pressure, lowers blood sugar and increases blood flow. This study will see if EGCG improves insulin resistance or insulin's effects on blood flow in people with insulin resistance.

Healthy normal weight or overweight people between 21 and 65 years of age may be eligible for this study. Participants are randomly assigned to take EGCG or a placebo ( inactive dummy pill ) in two 4-week treatment phases with a 2-week period of no study medication before each treatment phase. After the first 4-week treatment, patients on placebo are switched to EGCG and those on EGCG are switched to placebo. In addition to treatment, participants undergo the following procedures during the study period:

* Screening, including medical history, physical examination and blood and urine tests, and finger-stick blood sugar measurement for patients with diabetes
* Complete a dietary and physical activity questionnaire and consult with a dietitian
* Blood and urine tests
* At-home and clinic blood pressure monitoring
* Glucose clamp test to measure how the body responds to insulin. This test is done three times during the study. A needle is placed in a vein in each of the subject's arms, one for sampling blood and the other for infusing insulin, glucose and potassium. Glucose and insulin levels, electrolytes, lipids, fatty acids, cytokines and epicatechin are measured.
* Forearm blood flow measurement with microbubbles and ultrasound. Before beginning the glucose clamp test, a test of how well the blood vessels relax is done. A device that measures the size of the artery in the upper arm is placed above the elbow. Blood flow in the muscle of the forearm is measured by ultrasound using a small infusion through a vein of microbubble contrast agent consisting of gas-filled bubbles the size of red blood cells. The contrast agent is infused over a 7- to 9-minute period at the beginning of the glucose clamp test and again 2 hours after the beginning of the test.

DETAILED DESCRIPTION:
Green tea is a functional food whose consumption is associated with improved cardiovascular morbidity and mortality in several large epidemiological studies. One third of the solids in green tea are composed of the bioactive polyphenol epigallocatechin 3-gallate (EGCG). Studies in both cell- and animal-based models (from our lab and elsewhere) suggest that EGCG may mimic and/or augment beneficial metabolic, vascular, and anti-inflammatory actions of insulin. Indeed, we have recently shown that 3-week EGCG therapy of SHR rats (genetic model of hypertension with features of human metabolic syndrome including insulin resistance, hyperinsulinemia, endothelial dysfunction, and overweight) lowers blood pressure, improves endothelial dysfunction, increases insulin sensitivity, and raises adiponectin levels nearly as effectively as treatment with the conventional ACE-inhibitor enalapril. Obesity, type 2 diabetes, and hypertension are all important interrelated public health problems that are characterized by reciprocal relationships between insulin resistance and endothelial dysfunction. Thus, therapies for these diseases that improve insulin resistance often simultaneously improve endothelial function and vice versa. Based on results from cellular, physiological, and epidemiological studies, we hypothesize that oral EGCG administration will simultaneously ameliorate insulin resistance and lower blood pressure in human subjects with obesity. To test these hypotheses, we will conduct a randomized, placebo-controlled, double-blind, cross-over study to evaluate potential beneficial effects of EGCG to modulate insulin sensitivity, blood pressure, vascular function, and inflammatory markers in two groups of subjects (lean healthy controls, obesity). After a 2-week EGCG-free run-in period, each subject will be randomized to receive EGCG or placebo capsules (400 mg p.o. B.I.D.) for 4 weeks. This will be followed by a 2-week EGCG-free washout period after which subjects will cross-over to the other treatment arm. At baseline, and after each 4-week treatment period, we will assess insulin sensitivity (hyperinsulinemic isoglycemic glucose clamp technique) and vascular function. Regarding vascular function, we will measure basal and insulin-stimulated brachial artery blood flow (large conduit artery assessed by Doppler ultrasound) as well as capillary recruitment in forearm skeletal muscle (small nutritive arterioles assessed by ultrasound with microbubble contrast). Blood pressure will be measured weekly in the UMB GCRC throughout the duration of the study. EGCG pharmacokinetics will be measured at the beginning of each glucose clamp study day after oral administration of a single dose of EGCG or placebo. Finally, various plasma markers of inflammation will be measured at baseline and at the end of each treatment arm to evaluate potential changes that may be related to improvements in metabolic and/or vascular function. This study will explore whether EGCG, a single compound thought to be a major bioactive component of green tea, is effective at improving insulin resistance and lowering blood pressure in subjects with obesity. Results from this study may have important implications for understanding potential health benefits of functional foods that contain bioactive polyphenols including green tea, dark chocolate, and red wine.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY SUBJECTS:

Men and women in good general health with no significant underlying illnesses who are between the ages of 21-65 years of age with HbA(1C) less than 6.5%, fasting blood glucose less than 100 mg/dL, blood pressure less than 120/80, and BMI between 20-25 kg/m(2). Subjects should have never smoked tobacco or not smoked within the previous year.

OBESE SUBJECTS:

Men and women in good general health with no significant underlying illnesses except obesity who are between the ages of 21-65 years of age with HbA(1C) less than 6.5%, fasting blood glucose less than 110 mg/dl, blood pressure less than 140/90, and BMI between 30-40 kg/m(2).

EXCLUSION CRITERIA:

ALL SUBJECTS:

Subjects will be excluded from our study if they are pregnant , breastfeeding or if they plan pregnancy prior to the end of the study.

In addition, subjects will be excluded if their age is greater than 65 yrs, BMI greater than or equal to 40 kg/m(2), or have liver disease (including liver transaminase levels greater than twice the upper limit of normal), pulmonary disease, renal insufficiency (serum creatinine greater than 2.0 mg/dl), coronary heart disease, heart failure (New York Heart Association heart failure Class III or IV), peripheral vascular disease, coagulopathy, major depressive disorder, actively smoking or used tobacco within the last year, history of cancer, in treatment for any form of cancer, positive tests for HIV, hepatitis B or C, or take systemic corticosteroids, thiazolidinediones (within 3 months), insulin, or anticoagulants, use food supplements that cannot be discontinued, regular intake of 8 or more cups of tea per week within 3 months prior to study entry, regular alcoholic beverage intake of more than two drinks per day (a drink corresponds to approximately 12 ounces of beer, 4 ounces of table wine, and between 1 and 1.5 ounces of 80-proof spirits), poor compliance during run-in period or regular use of medications that affect insulin sensitivity, blood pressure or vascular function and that cannot be discontinued.

In addition, history of any other medical disease, laboratory abnormalities, or psychological conditions that would make the subject (based upon the principal investigator's judgment) unsuitable for study enrollment.

Subjects with known hypersensitivity to octafluoropropane, recent eye surgery, or with known cardiac shunts will also be excluded from participating because of potential adverse effects from microbubble contrast agent.

Subjects will be excluded if they are unable to give informed consent for all procedures.

Currently, type 2 diabetes is not rare in children, however children are excluded from this study because children do not typically take EGCG and do not typically have hypertension or type 2 diabetes mellitus.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement in insulin resistance | 14 weeks
  measurements of insulin resistance prior to study drug, after 4 weeks of EGCG or placebo and at end of study

SECONDARY OUTCOMES:
Improvement in endothelial dysfunction | 14 weeks
  measurements of endothelial function prior to study drug, after 4 weeks of EGCG or placebo and at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Munir, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Jemal A, Ward E, Hao Y, Thun M. Trends in the leading causes of death in the United States, 1970-2002. JAMA. 2005 Sep 14;294(10):1255-9. doi: 10.1001/jama.294.10.1255. PMID 16160134
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Fox CS, Coady S, Sorlie PD, Levy D, Meigs JB, D'Agostino RB Sr, Wilson PW, Savage PJ. Trends in cardiovascular complications of diabetes. JAMA. 2004 Nov 24;292(20):2495-9. doi: 10.1001/jama.292.20.2495. PMID 15562129